CLINICAL TRIAL: NCT00041080
Title: A Randomized Study Of Tamoxifen Versus Thalidomide (NSC# 66847) In Patients With Biochemical-Recurrence-Only Epithelial Ovarian Cancer, Cancer Of The Fallopian Tube, And Primary Peritoneal Carcinoma After First Line Chemotherapy
Brief Title: Tamoxifen Compared With Thalidomide in Treating Women With Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02475; NCI-2012-02475 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000069441; GOG-0198 (Other: Gynecologic Oncology Group); GOG-0198 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Fallopian Tube Cancer; Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer; Stage III Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Tamoxifen; Thalidomide

ARMS (2):
- Arm I (thalidomide) (Experimental): Patients receive oral thalidomide once daily on days 1-28.
  Interventions: Drug: thalidomide; Other: laboratory biomarker analysis
- Arm II (tamoxifen) (Experimental): Patients receive oral tamoxifen twice daily on days 1-28.
  Interventions: Drug: tamoxifen citrate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tamoxifen citrate — Given orally
  Other Names: Nolvadex; TAM; tamoxifen; TMX
  Arms: Arm II (tamoxifen)
Drug: thalidomide — Given orally
  Other Names: Kevadon; Synovir; THAL; Thalomid
  Arms: Arm I (thalidomide)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Randomized phase III trial to compare the effectiveness of tamoxifen with that of thalidomide in treating women who have recurrent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer. Estrogen can stimulate the growth of some types of cancer cells. Hormone therapy using tamoxifen may fight cancer by blocking the uptake of estrogen. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. It is not yet known whether thalidomide is more effective than tamoxifen in treating ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the recurrence-free survival of women receiving tamoxifen or thalidomide for epithelial ovarian cancer, cancer of the fallopian tube, or primary peritoneal carcinoma who are in complete clinical remission following front-line treatment but have a high risk of recurrence due to rising serum CA-125.

II. To compare the toxicities and complications of these treatments.

SECONDARY OBJECTIVES:

I. To determine whether changes in serum biomarker levels including VEGF and/or bFGF are independent of the randomization treatment.

II. To determine whether serum and plasma biomarker levels including VEGF and/or bFGF are associated with the duration of recurrence-free survival.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to the interval between completion of front-line chemotherapy and appearance of biochemical progression (6 months or less vs more than 6 months). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral thalidomide once daily on days 1-28.

ARM II: Patients receive oral tamoxifen twice daily on days 1-28.

In both arms, courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients may receive additional therapy beyond 1 year at the investigator's discretion.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage III or IV ovarian epithelial, fallopian tube, or primary peritoneal cancer that was treated with only 1 prior first-line chemotherapy regimen (platinum/taxane-based)
* Clinically and radiologically without evidence of measurable and nonmeasurable disease

  * Symptomatic ascites and pleural effusions are considered nonmeasurable disease
* Must have a biochemical recurrence

  * CA 125 must have been normal prior to or normalized during first-line therapy and then subsequently rose to exceed twice the upper limit of normal
  * Patients entering study with a CA 125 level less than 100 U/mL must be confirmed a second time within a period of not more than 4 weeks
  * Patients with a CA 125 level of at least 100 U/mL may be entered without confirmatory measurement
* Ineligible for a higher priority Gynecologic Oncology Group protocol (if one exists)
* No history of brain metastases
* Performance status - GOG 0-1
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 60 mL/min
* No history of deep venous thrombosis
* No prior cerebrovascular accident
* No history of pulmonary embolism
* No significant infection
* No grade 2 or greater sensory or motor neuropathy
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use at least 1 highly active method and at least 1 additional effective method of contraception for 4 weeks before, during, and for 4 weeks after study participation
* No prior immunotherapy (e.g., interleukins)
* No prior biological response modifiers (e.g., monoclonal antibodies)
* No prior antiangiogenic agents (e.g., carbonic anhydrase inhibitors)
* At least 3 weeks since prior anticancer chemotherapy and recovered
* No prior or concurrent tamoxifen or other selective estrogen receptor modulators
* At least 4 weeks since prior and no concurrent hormones (e.g., estrogen or progesterone)
* At least 3 weeks since prior anticancer radiotherapy and recovered
* At least 3 weeks since prior anticancer surgery and recovered
* Prior second-look surgery without cytoreduction allowed
* At least 3 weeks since other prior anticancer therapy and recovered
* No prior interval cytoreduction
* No concurrent full-dose therapeutic anticoagulation
* No concurrent antiseizure medications for seizure disorder
* No concurrent bisphosphonates (e.g., zoledronate)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2003-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Hurteau, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began Feb 3, 2003 and completed Jan 30, 2011. All patients were enrolled from GOG member institutions in the United States.
Pre-assignment Details: Eligible patients had histologically confirmed ovarian, fallopian tube or primary peritoneal cancer. They had rising CA-125 that exceeded twice the upper-limit of normal, but no radiographic or physical evidence of disease following first-line chemotherapy.
Groups:
- Grp - 1: Thalidomide 200mg orally daily with weekly escalation of 100mg to a maximum dose of 400mg until progression or additional therapy prohibited further therapy.
- Grp - 2: Tamoxifen 20mg orally twice daily for up to 12 28-day cycles until progression or adverse effect prohibited additional therapy.
Period: Overall Study
Arm/Group | Grp - 1 | Grp - 2
Started | 69 (number patients enrolled on study) | 70 (number patients enrolled on study)
Completed | 39 | 60
Not Completed | 30 | 10
Not completed — Adverse Event | 21 | 1
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Concommitant Illness/Other | 1 | 2
Not completed — Did not start therapy | 1 | 1
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: Description of population is based on eligible patients.
  1 patient not included in characteristics due to ineligible primary tumor site.
Groups:
- Grp - 2: Tamoxifen 20mg orally for up to 12 28-day cycles until progression or adverse effect prohibited additional therapy.
- Total: Total of all reporting groups
Arm/Group | Grp - 1 | Grp - 2 | Total
Number analyzed (Participants) | 68 | 70 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.8) | 61.6 (10.5) | 62.9 (10.7)
Age, Customized [Number; unit: participants]
  < 50 years | 7 | 12 | 19
  50-59 years | 17 | 14 | 31
  60-69 years | 22 | 28 | 50
  70-79 years | 17 | 15 | 32
  80-89 years | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 70 | 138
  Male | 0 | 0 | 0
Gynecologic Oncology Group (GOG) Performance Status [Number; unit: participants]
  0 - asymptomatic | 63 | 67 | 130
  1 - symptomatic | 5 | 3 | 8
Primary Site of Disease [Number; unit: participants]
  Ovary | 58 | 59 | 117
  Peritoneum | 10 | 10 | 20
  Fallopian Tube | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival
Time Frame: from enrollment onto the study until first disease progression or death due to any cause
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Grp - 1 | Grp - 2
Number analyzed (Participants) | 68 | 70
months | 3.2 [2.7 to 3.9] | 4.5 [2.7 to 5.5]

ADVERSE EVENTS:
Time Frame: Within 30 days after stopping study treatment or any SAE that the study investigator felt was study treatment related.
Description: Other Adverse Events(AEs) are at least possibly related to study treatment. Due to the methods in which adverse events were collected and/or stored for this study, it is not possible to report only the Other (not including Serious) AEs in the appropriate table. Therefore, the Other AEs table includes a combined set of serious and non-serious AEs.
Arm/Group | Grp - 1 | Grp - 2
Serious Adverse Events (participants affected / at risk) | 3/67 | 1/69
Other Adverse Events (participants affected / at risk) | 42/67 | 24/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Grp - 1 (N=67) | Grp - 2 (N=69)
Neutropenia/Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Thrombosis/embolism (Cardiac disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Partial small bowel obstruction (Gastrointestinal disorders) | 1 | 0
SGPT (Hepatobiliary disorders) | 1 | 0
Febrile Neutropenia (Infections and infestations) | 1 | 0
Edema (Blood and lymphatic system disorders) | 1 | 0
Neuropathy - motor (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Dizziness/lightheadedness (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Grp - 1 (N=67) | Grp - 2 (N=69)
Leukopenia (Blood and lymphatic system disorders) | 25 | 8
Neutropenia (Blood and lymphatic system disorders) | 21 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4
Anemia (Blood and lymphatic system disorders) | 15 | 10
DVT/thrombosis (Cardiac disorders) | 4 | 1
Other cardiovascular (Cardiac disorders) | 11 | 6
Constitutional (General disorders) | 42 | 18
Dermatologic (Skin and subcutaneous tissue disorders) | 22 | 4
Endocrine (Endocrine disorders) | 1 | 24
Gastrointestinal (Gastrointestinal disorders) | 42 | 22
Genitourinary/renal (Reproductive system and breast disorders) | 3 | 5
Metabolic (Metabolism and nutrition disorders) | 8 | 8
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 | 4
Somnolence (Nervous system disorders) | 17 | 0
Other neurologic (Nervous system disorders) | 32 | 2
Peripheral neurologic (Nervous system disorders) | 32 | 9
Ocular/visual (Eye disorders) | 11 | 2
Pain (General disorders) | 26 | 19
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 11 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less